CLINICAL TRIAL: NCT05240287
Title: Evaluation Of Balance, Plantar Pressure Distribution and Gait in Adults With Pes Planus
Brief Title: Balance, Plantar Pressure Distribution and Gait in Pes Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ozlem Yuruk, Assoc. Prof., Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: KA21/410
Record Dates: First submitted 2021-11-20; First posted 2022-02-15 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Pes Planus
Keywords: pes planus; balance; gait
MeSH Terms: conditions — Flatfoot | interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group -adults with pes planus (Active Comparator): * Individuals between the ages of 20-45
  * Individuals with bilateral pes planus according to the Navicular Drop Test and Foot Posture Index
  Interventions: Diagnostic Test: Navicular Drop Test; Diagnostic Test: Foot Posture Index; Diagnostic Test: Balance; Diagnostic Test: Plantar Pressure Analysis; Diagnostic Test: Gait Analysis
- Control group -adults without pes planus (normal foot) (Other): * Individuals between the ages of 20-45
  * Individuals without pes planus according to the Navicular Drop Test and Foot Posture Index
  Interventions: Diagnostic Test: Navicular Drop Test; Diagnostic Test: Foot Posture Index; Diagnostic Test: Balance; Diagnostic Test: Plantar Pressure Analysis; Diagnostic Test: Gait Analysis

INTERVENTIONS:
Diagnostic Test: Navicular Drop Test — The researchers will measure the distance between the navicular tuberosity and the ground with a caliper with non-weight bearing in sitting. After that, the distance between the ground and the navicular tuberosity will be measured in standing while weight-bearing. The researchers will evaluate both sides and record the value in mm. According to Navicular Drop Test, the difference between weighted and unweighted measurements is considered normal (neutral) if it is between 5 and 9 mm, pronation (pes planus) if it is 10 mm or more, and supination (pes cavus) if it is 4 mm or less. In our study, individuals with a difference of 10 mm or more in both feet will be included in the pes planus, and individuals with a difference between 5-9 mm will be included in the control group.
Diagnostic Test: Foot Posture Index — The index consists of six items in which the foot is evaluated observationally. In the evaluation, the individual is asked to stand in a comfortable and relaxed position. The researcher observes the medial longitudinal arch structure, the structure of the talonavicular joint region, the degree of abduction/adduction in the forefoot relative to the hindfoot in the front part of the foot. In the back foot, inversion/eversion of the calcaneus, talus head position, and curvatures above and below the lateral malleolus are evaluated. The total score is reached by scoring each criterion between -2 and +2 values. 0; neutral position, (+) values; pronation (pes planus), (-) values indicate supination (pes cavus). Individuals with +6 to +12 points from this index will be included in our study.
Diagnostic Test: Balance — Static and dynamic balance and stability limit values of individuals will be evaluated with the HUR Smart Balance (SME Inc, USA) balance measurement device. The device consists of a computer and a platform on which individuals can place their feet. For static balance measurement, individuals will be asked to place their feet on the marked places on the platform. The researchers will evaluate the balance in four different situations, 30 seconds each. In the first test, individuals keep the balance on firm ground with their eyes open. The second test performed on the firm ground with eyes closed, in the third test, on the soft ground with eyes open, and in the fourth test, on the soft ground with eyes closed. For dynamic balance, individuals will be asked to extend their body weight to the front, back, and sides with their feet in 4 different directions for 8 seconds.
Diagnostic Test: Plantar Pressure Analysis — Plantar pressure analysis of individuals will be evaluated by measuring with the DIERS Pedoscan DICAM 3 v3.10.8 (2019) device. DIERS Pedoscan is a system integrated into the treadmill that measures the pressure distribution on the sole during stance. As a result of this evaluation, right-left and anterior-posterior weight transfer, left-right foot rotation, lateral mobility, the center of gravity movement, and swing area data will be recorded.
Diagnostic Test: Gait Analysis — Gait analysis of individuals will be evaluated with the DIERS Leg Axis DICAM 3 v3.10.8 (2019) system. The system consists of a treadmill, computer, and cameras. Before the measurement, colored markers will be placed on the knee and ankle joints of the individual. For gait assessment, individuals will walk at their preferred comfortable walking speed. In the evaluation, joint angles, walking speed, step lengths are recorded. Evaluation time is approximately 5 minutes.

SUMMARY:
Introduction:The results of studies evaluating balance, plantar pressure analysis, and gait in adults with pes planus have differed in the literature. The aim of this study is to evaluate balance, plantar pressure, and gait in adults with pes planus and compare them with adults without pes planus.

Materials and Methods: The study will be conducted at the Ministry of Youth and Sports, Athletic Training and Research Center. A total of 118 individuals, 59 individuals with pes planus and 59 individuals without pes planus, will be included in the study according to the Navicular Drop Test and Foot Posture Index. In the study, the descriptive characteristics of the individuals will be recorded. Static and dynamic balance measurements, plantar pressure analysis and gait analysis of individuals will be performed, and the two groups will be compared.

Results: The data will be analyzed using the statistical program for social sciences (SPSS) version 21.0 (IBM SPSS Statistics for Windows, Armonk, NY: IBM Corp.). The data will be expressed as mean standard deviation (X±SD) and number (n%). The homogeneity of the groups will be evaluated with the Levene Test. Balance, plantar pressure, and walking values between the groups will be compared using the "Mann Whitney-U" Test. All the statistical analyses will be set a priori at an alpha level of p<0.05.

Discussion: The results will be discussed in the light of the recent literature. In the literature, there are conflicting results about the balance and gait of adults with pes planus. The study can contribute to the literature in this respect.

DETAILED DESCRIPTION:
Introduction The lower extremity kinematic chain includes foot, ankle, knee, and hip joints. The foot is a complex structure and provides the body's contact with the ground. The foot is one of the most important sources of somatosensory information required for balance and walking. The proprioceptive information from the joints, muscles, and ligaments of the foot maintains the upright posture. Also, it helps to absorb ground reaction forces during walking and provides balance by adapting to different grounds.

The arches of the foot have a critical role in stability and flexibility. These arches have functions such as carrying body weight, contributing to the gait cycle, and generating energy. The foot has two longitudinal arches in the transverse plane: the medial longitudinal arch and the lateral longitudinal arch. The calcaneus, talus, navicular, cuneiform I, II, III, and the first three metatarsal bones form the medial longitudinal arch. The arch is the primary weight-bearing and shock-absorbing structure of the foot. The talonavicular joint, the subtalar joint, and the tibialis posterior muscle protect the structure of this arch.

Pes planus is defined as the decrease or complete disappearance of the medial longitudinal arch of the foot. It is the most common deformity among foot deformities. All babies have pes planus on their feet from birth. The medial longitudinal arch may not form in the feet of healthy infants until the age of 3 years. In advancing age, the development of the midtarsal joints and bones is supported by the strengthening of the ligaments, and the medial arch develops. However, with the weakness of the plantar fascia and muscle groups that support the medial longitudinal arch, arch support may decrease, and pes planus may be seen. In addition, it can be seen as a result of excessive load on the plantar fascia in adults who stand on hard floors for a long time due to their profession, in obese individuals, in cases with muscle imbalance, or as a result of the progression of pes planus in childhood. In a study on pes planus and pes cavus; 60% of the population had a normal foot structure, while 20% had a pes planus foot structure, and 20% had a pes cavus foot structure.

Pes planus causes a change in the load distribution in the medial side of the foot. The number of loads on the lower extremity joints and lumbar vertebrae vary. Various symptoms are seen after this biomechanical change. The symptoms are pain, loss of strength, fatigue, instability, and functional limitations, especially with walking and standing. As a result of the energy expenditure of the individuals during gait also increases. The increased energy expenditure negatively affects lower extremity performance .

Balance is the ability to keep the body's center of gravity within the acceptable limits of the support surface during activities such as sitting, standing, or gait. Balance is a complex process involving multifaceted sensory, motor, and biomechanical components. It is divided into two as static and dynamic balance. Changes in the normal alignment of the foot in pes planus cause abnormal sensory input from the foot, which prevents proper muscle activity required for posture and postural swings. This condition may cause balance problems. While some studies in the literature have shown that static postural stability, which is evaluated by force plate or balance systems, decreases in individuals with pes planus, others reported no difference compared to the neutral foot. Kim et al. stated that static stability is better in individuals with pes planus than in individuals without pes planus. The authors also found that there was no difference in dynamic stability. Plantar pressure distribution is a factor that affects both balance and gait. It has been observed that individuals with pes planus give more weight to the big toe, middle of the forefoot, and medial foot compared to the neutral foot. However, in another study, the same researchers compared pes planus, pes cavus, and foot pressure center in normal feet and found that only the terminal phase of the stance and the pre-swing phase differed. Although some evidence of characteristic plantar pressure patterns has been identified, differences in gait analysis protocols and plantar pressure analysis techniques make it difficult to obtain a clear result.

The gait cycle is affected by many pathologies. Some factors such as deformities, loss of muscle strength, decreased motor or sensory control, balance problems adversely affect the gait cycle and cause gait disturbance. As a result, compensatory movements occur. Pes planus may also affect the gait cycle. It has been found that pes planus can cause the foot to go pronation and plantar flexion, adduction of the talus, and valgus of the calcaneus during load-bearing to the extremity. Hunt et al. performed a kinetic and kinematic analysis in the stance phase of walking in individuals with pes planus. However, the investigators found no difference between individuals with pes planus and the control group. The investigators stated that this result was due to the mild and asymptomatic pes planus of the individuals.

All these biomechanical problems can lead to metatarsal stress fractures, plantar fasciitis, Achilles tendonitis, tibialis anterior inflammation, or patellofemoral joint pain in the long term. For this reason, it is necessary to evaluate pes planus from multiple perspectives and to recommend appropriate treatment approaches.

As can be seen, the results of studies evaluating balance, plantar pressure analysis, and gait in adults with pes planus have differed in the literature. In addition, studies using objective computerized systems are few. The aim of this study is to evaluate balance, plantar pressure, and gait in adults with pes planus and compare them with adults without pes planus.

Hypothesis 1:There is no difference between the static and dynamic balance values of adults with pes planus and without pes planus.

Hypothesis 2:There is no difference between the plantar pressure distribution values of adults with pes planus and without pes planus.

Hypothesis 3:There is no difference between the gait parameters of adults with pes planus and without pes planus.

Methods Participants

The university students and workers in Baskent University who meet the inclusion criteria will be contacted and invited to study. There will be two groups in the study:

Study group -adults with pes planus Control group -adults without pes planus (normal foot) For the sample size calculation G*Power Ver. 3.0.10 (Franz Faul, Universität Kiel, Germany) was used. The sample size of the study was calculated with 85% power and 0.05 margin of error, and it was found that a total of 118 individuals, 59 individuals in each group, should be included in the study.

Method In the study, the descriptive characteristics of the participants will be recorded. Then, by applying the Navicular Drop Test and the Foot Posture Index, participants will be divided into two groups as those with pes planus and those without pes planus.

Navicular Drop Test The navicular drop test is one of the static foot assessment tool. The researchers will measure the distance between the navicular tuberosity and the ground with a caliper with non-weight bearing in sitting. After that, the distance between the ground and the navicular tuberosity will be measured in standing while weight-bearing. The researchers will evaluate both sides and record the value in mm. According to Navicular Drop Test, the difference between weighted and unweighted measurements is considered normal (neutral) if it is between 5 and 9 mm, pronation (pes planus) if it is 10 mm or more, and supination (pes cavus) if it is 4 mm or less. In the study, individuals with a difference of 10 mm or more in both feet will be included in the pes planus, and individuals with a difference between 5-9 mm will be included in the control group.

Foot Posture Index The index consists of six items in which the foot is evaluated observationally. In the evaluation, the individual is asked to stand in a comfortable and relaxed position. The researcher observes the medial longitudinal arch structure, the structure of the talonavicular joint region, the degree of abduction/adduction in the forefoot relative to the hindfoot in the front part of the foot. In the back foot, inversion/eversion of the calcaneus, talus head position, and curvatures above and below the lateral malleolus are evaluated. The total score is reached by scoring each criterion between -2 and +2 values. 0; neutral position, (+) values; pronation (pes planus), (-) values indicate supination (pes cavus). Individuals with +6 to +12 points from this index will be included in the study. Since this index is an evaluator-based scale, no Turkish validity study has been conducted.

Balance Static and dynamic balance and stability limit values of individuals will be evaluated with the HUR Smart Balance (SME Inc, USA) balance measurement device. The device consists of a computer and a platform on which individuals can place their feet. For static balance measurement, individuals will be asked to place their feet on the marked places on the platform. The researchers will evaluate the balance in four different situations, 30 seconds each. In the first test, individuals keep the balance on firm ground with their eyes open. The second test performed on the firm ground with eyes closed, in the third test, on the soft ground with eyes open, and in the fourth test, on the soft ground with eyes closed. For dynamic balance, individuals will be asked to extend their body weight to the front, back, and sides with their feet in 4 different directions for 8 seconds and reach the last point where the sole does not break with the ground. The device gives the balance value as a printout by calculating the deviation rate of the individual from the target and the risk of falling forward, backward, and sideways. The measurement takes an average of 10 minutes.

Plantar Pressure Analysis Plantar pressure analysis of individuals will be evaluated by measuring with the DIERS Pedoscan DICAM 3 v3.10.8 (2019) device. DIERS Pedoscan is a system integrated into the treadmill that measures the pressure distribution on the sole during stance. As a result of this evaluation, right-left and anterior-posterior weight transfer, left-right foot rotation, lateral mobility, the center of gravity movement, and swing area data will be recorded.

Gait Analysis Gait analysis of individuals will be evaluated with the DIERS Leg Axis DICAM 3 v3.10.8 (2019) system. The system consists of a treadmill, computer, and cameras. Before the measurement, colored markers will be placed on the knee and ankle joints of the individual. For gait assessment, individuals will walk at their preferred comfortable walking speed. In the evaluation, joint angles, walking speed, step lengths are recorded. Evaluation time is approximately 5 minutes.

Statistical analysis The data will be analyzed using the statistical program for social sciences (SPSS) version 21.0 (IBM SPSS Statistics for Windows, Armonk, NY: IBM Corp.). The data will be expressed as mean standard deviation (X±SD) and number (n%). The homogeneity of the groups will be evaluated with the Levene Test. Balance, plantar pressure, and walking values between the groups will be compared using the "Mann Whitney-U" Test. All the statistical analyses will be set a priori at an alpha level of p<0.05.

Importance of the study In this study, researchers will expect that the balance, plantar pressure distribution, and gait parameters of adults with pes planus are different from healthy individuals. In the literature, there are conflicting results about the balance and gait of adults with pes planus. The researchers think that the study will contribute to the literature in this respect.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria of individuals with pes planus:

* Individuals between the ages of 20-45
* Individuals with bilateral pes planus according to the Navicular Drop Test and Foot Posture Index

Inclusion criteria for individuals without pes planus:

* Individuals between the ages of 20-45
* Individuals without pes planus according to the Navicular Drop Test and Foot Posture Index

Exclusion Criteria:

* Individuals who had trauma, fall, injury in the last six months
* Individuals who have a chronic disease that affects gait and balance
* Individuals who have had lower extremity surgery
* Individuals who received any medical treatment during the study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Static and Dynamic Balance | 10 minutes
  Balance is the ability to keep the body's center of gravity within the acceptable limits of the support surface during activities such as sitting, standing, or gait. Static and dynamic balance and stability limit values of individuals will be evaluated with the HUR Smart Balance (SME Inc, USA) balance measurement device.

SECONDARY OUTCOMES:
Plantar Pressure Analysis-weight transfer | 5 minutes
  Plantar pressure analysis of individuals will be evaluated by measuring with the DIERS Pedoscan DICAM 3 v3.10.8 (2019) device. DIERS Pedoscan is a system integrated into the treadmill that measures the pressure distribution on the sole during stance. As a result of this evaluation, right-left and anterior-posterior weight transfer will be recorded as milimeters.
Plantar Pressure Analysis- left-right foot rotation | 5 minutes
  Plantar pressure analysis of individuals will be evaluated by measuring with the DIERS Pedoscan DICAM 3 v3.10.8 (2019) device. DIERS Pedoscan is a system integrated into the treadmill that measures the pressure distribution on the sole during stance. As a result of this evaluation, left-right foot rotation will be recorded as milimeters.
Plantar Pressure Analysis- the center of gravity movement | 5 minutes
  Plantar pressure analysis of individuals will be evaluated by measuring with the DIERS Pedoscan DICAM 3 v3.10.8 (2019) device. DIERS Pedoscan is a system integrated into the treadmill that measures the pressure distribution on the sole during stance. As a result of this evaluation the center of gravity movement will be recorded as milimeters.
Plantar Pressure Analysis- swing area | 5 minutes
  Plantar pressure analysis of individuals will be evaluated by measuring with the DIERS Pedoscan DICAM 3 v3.10.8 (2019) device. DIERS Pedoscan is a system integrated into the treadmill that measures the pressure distribution on the sole during stance. As a result of this evaluation swing area data will be recorded as mm2
Gait analysis-Joint angles | 5 minutes
  Gait analysis of individuals will be evaluated with the DIERS Leg Axis DICAM 3 v3.10.8 (2019) system. The system consists of a treadmill, computer, and cameras. Before the measurement, colored markers will be placed on the knee and ankle joints of the individual. For gait assessment, individuals will walk at their preferred comfortable walking speed. In the evaluation hip, knee and ankle joint angles will be recorded as degree
Gait analysis-walking speed | 5 minutes
  Gait analysis of individuals will be evaluated with the DIERS Leg Axis DICAM 3 v3.10.8 (2019) system. The system consists of a treadmill, computer, and cameras. Before the measurement, colored markers will be placed on the knee and ankle joints of the individual. For gait assessment, individuals will walk at their preferred comfortable walking speed. In the evaluation walking speed will be recorded as meter/second.
Gait analysis- step lengths | 5 minutes
  Gait analysis of individuals will be evaluated with the DIERS Leg Axis DICAM 3 v3.10.8 (2019) system. The system consists of a treadmill, computer, and cameras. Before the measurement, colored markers will be placed on the knee and ankle joints of the individual. For gait assessment, individuals will walk at their preferred comfortable walking speed. In the evaluation step lengths will be recorded as centimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Yasin Acar, PT, Study Chair — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No